CLINICAL TRIAL: NCT00507871
Title: Prevalence and Clinical Presentation of Respiratory Cryptosporidiosis Among Children With Diarrhea in Mulago Hospital, Uganda
Brief Title: Transmission and the Respiratory Tract in Cryptosporidiosis
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jeffrey K Griffiths, Associate Professor, Tufts University School of Medicine
Other Study IDs: 06-0033
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2007-09

CONDITIONS: Cryptosporidiosis
Keywords: cryptosporidiosis, Cryptosporidium, Uganda, diarrhea
MeSH Terms: conditions — Cryptosporidiosis; Diarrhea

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Cryptosporidium is an intestinal parasite that causes diarrhea in children and adults. In addition to infection of the stomach, this parasite can infect the respiratory system causing a cough and/or problems breathing. This study will enroll 480 children between the ages of 9 and 36 months who come to Mulago Hospital for treatment of diarrhea. Researchers believe a large number of children with diarrhea and cough will have the parasite present in their sputum (mucus coughed up). Researchers also believe that children who have respiratory tract cryptosporidiosis may have a cough, increased number of breaths per minute, and/or a lower oxygen level. Blood, stool, saliva, and sputum samples will be collected from all children in the study and tested for Cryptosporidium. Children too young to provide a sputum sample will have a tube placed to collect a mucus sample from the lungs. Study participation may be as short as 4 hours or as long as 2 days depending on each child's health.

DETAILED DESCRIPTION:
Cryptosporidiosis is recognized as a major cause of diarrhea worldwide. In addition to infection of the gastrointestinal tract and associated fecal-oral transmission, there is evidence that Cryptosporidium can infect the respiratory tract. Of particular interest are numerous reports indicating that respiratory symptoms occur with considerable frequency in subjects with intestinal cryptosporidiosis although the etiology of the respiratory symptoms was never investigated. The association between respiratory symptoms and intestinal cryptosporidiosis is particularly strong in children with questionable nutritional status. This study will evaluate the prevalence and clinical presentation of respiratory cryptosporidiosis among children with diarrhea in Mulago Hospital, Kampala, Uganda. The study will screen approximately 1536 children aged 9-36 months who present to the Acute Care Unit of Mulago Hospital in Kampala, Uganda, with acute or persistent diarrhea. Based on the results of fecal testing, 480 children will be actively selected to undergo further sample collection in 2 groups. Group 1 will be comprised of children with Cryptosporidium-positive stools, approximately 50% of whom are expected to have cough (n=384). Group 2 will be comprised of children with Cryptosporidium-negative stools and cough (n=96). The primary objectives of the study are: to establish the prevalence of cough in children with diarrhea due to Cryptosporidium infection; to establish the prevalence of respiratory tract cryptosporidiosis in children with diarrhea due to Cryptosporidium infection; to establish the prevalence of respiratory tract cryptosporidiosis in children with diarrhea due to other causes; and to determine whether respiratory Cryptosporidium infection in children is associated with increased respiratory rates and decreased oxygen saturation levels. To address these objectives, the study will focus on whether Cryptosporidium oocysts can be recovered from induced sputum of subjects who have acute or persistent diarrhea and are concurrently experiencing a cough or unexplained tachypnea or hypoxemia. The primary clinical measures include: duration of diarrhea (days); presence and duration of cough (days); respiratory rate at presentation and if dehydrated, after rehydration; oxygen saturation (as measured by pulse oximetry) at presentation; and oxygen therapy requirement and oxygen saturation after 30 minutes of oxygen therapy if initial saturation is <92%. Primary parasitological measures include: presence or absence of Cryptosporidium in stool (as detected by modified acid fast staining and PCR); presence or absence of Cryptosporidium in sputum (as detected by PCR); and presence or absence of Cryptosporidium in saliva (as detected by PCR). Secondary clinical measures include: HIV status (determined by voluntary HIV testing via enzyme-linked immunosorbent assay + reverse transcriptase PCR in children aged less than 18 months); CD4+ counts/percentages (as measured by flow cytometry in children tested for HIV); concurrent respiratory infection (as determined by processing of sputum for routine bacterial pathogens, tuberculosis and pneumocystis jirovecii pneumonia; anemia (determined by hemoglobin measurement from complete blood count); and nutritional status (as determined from the weight-for-age score, height-for-age score, weight-for-height score, head circumference, and mid upper arm circumference). Secondary parasitological measurements include: species of Cryptosporidium in stool, in sputum, and in saliva (as determined by restriction fragment length polymorphism). Subject participation duration in the study is dependent on the health status of the child at admission and the extent of clinical care required. In uncomplicated cases, subject duration may be as short as 4 hours. In subjects requiring extensive clinical care subject duration may extend to 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 9-36 months at the time of enrollment
* Presence of acute or persistent diarrhea (diarrhea defined as 3 or more loose stool in the previous 24 hours AND not considered normal for that child if the child is exclusively breast fed OR any number of bloody stools in the previous 24 hours; less than or equal to 14 days duration for acute diarrhea; >14 days duration for persistent diarrhea)
* Child's parent/guardian speaks English or Luganda
* Parent/guardian provides full and free informed consent for child to participate in study

Exclusion Criteria:

* Unknown age
* Known cardiac, CNS, metabolic or endocrine disorders
* Moribund children
* Children with recent history of choking or sudden onset of symptoms with suspected foreign body inhalation

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children attending the Acute Care Unit at Mulago Hospital, Kampala, Uganda
Sampling Method: Non-Probability Sample
Enrollment: 480
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrery K Griffiths, MD, Principal Investigator — Tufts Universtiy
Locations (1):
- Makerere University Medical School, Kampala, Uganda

REFERENCES:
- [Derived] Mor SM, Tumwine JK, Ndeezi G, Srinivasan MG, Kaddu-Mulindwa DH, Tzipori S, Griffiths JK. Respiratory cryptosporidiosis in HIV-seronegative children in Uganda: potential for respiratory transmission. Clin Infect Dis. 2010 May 15;50(10):1366-72. doi: 10.1086/652140. PMID 20377408